CLINICAL TRIAL: NCT01991860
Title: Randomized, Double-blind, Placebo-controlled Phase III Study of APD421 (Amisulpride for IV Injection) as Prophylaxis Against Post-operative Nausea and Vomiting
Brief Title: US Phase III Study of APD421 in PONV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Acacia Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DP10015
Record Dates: First submitted 2013-11-11; First posted 2013-11-25 (Estimated); Results first posted 2018-09-06 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-01

CONDITIONS: PONV
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Injections, Intravenous; Amisulpride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- APD421 (Experimental): APD421 (amisulpride), at 5mg given by single intravenous (IV) administration by slow push over one minute at induction of anaesthesia.
  Interventions: Drug: APD421- Amisulpride for IV injection
- Placebo (Placebo Comparator): Matching placebo given by single IV administration by slow push over one minute at induction of anaesthesia
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: APD421- Amisulpride for IV injection — APD421 ( Amisulpride) at 5mg given by single intravenous (IV) administration, by slow push over one minute, at induction of anaesthesia
  Other Names: Amisulpride for IV injection
  Arms: APD421
Drug: Placebo — Matching Placebo given by single intravenous (IV) administration, by slow push over one minute, at induction of anaesthesia
  Arms: Placebo

SUMMARY:
A comparison of the efficacy of APD421 and placebo in the prevention of PONV in patients at moderate-to-high risk of PONV.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age
* Patients undergoing elective surgery (open or laparoscopic technique) under general anaesthesia, expected to last at least one hour from induction of anaesthesia to wound closure and expected to require at least one overnight stay in hospital

Exclusion Criteria:

* Patients scheduled for outpatient/day case surgery
* Patients scheduled to undergo intra-thoracic, transplant or central nervous system surgery
* Patients scheduled to receive only a local anaesthetic/regional neuraxial (intrathecal or epidural) block
* Patients who are expected to remain ventilated for a period after surgery
* Patients who are expected to need a naso- or orogastric tube in situ after surgery is completed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2013-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tong J Gan, MD, Principal Investigator — Duke University Medical College
Locations (1):
- Duke, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 364 patients enrolled in the study (i.e. signed informed consent form), 22 patients were not randomised and not dosed. Of these, 4 withdrew their consent, 3 did not comply with the protocol procedures and 15 were not dosed for other unspecified reasons.
Groups:
- 5mg APD421: A 5mg (2mL) dose of APD421 given by slow intravenous (IV) push over one minute at induction of anaesthesia
- Placebo: 2mL of placebo given by slow intravenous (IV) push over one minute at induction of anaesthesia
Period: Overall Study
Arm/Group | 5mg APD421 | Placebo
Started | 176 | 166
Completed | 172 | 164
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Population: A total of 342 patients were randomised and dosed, comprising 176 randomised to APD421 and 166 to placebo. Of these, 4 patients from the APD421 group and 2 patients from the placebo group discontinued prematurely after randomisation
Groups:
- 5mg Dose APD421: A 5mg dose of APD421 given by slow push, single intravenous (IV) administration over a time frame of one minute at induction of anaesthesia
- Placebo: Single dose placebo given through intravenous (IV) administration
- Total: Total of all reporting groups
Arm/Group | 5mg Dose APD421 | Placebo | Total
Number analyzed (Participants) | 176 | 166 | 342
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.5 (14.2) | 53.0 (13.7) | 53.8 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 110 | 224
  Male | 62 | 56 | 118
Region of Enrollment [Number; unit: participants]
  United States | 176 | 166 | 342

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response
Description: The primary efficacy analysis was a comparison of the incidence of Complete Response, defined as no emesis (vomiting or retching) and no use of rescue medication in the 24 hours after the end of surgery, between the active group and the placebo group using Pearson χ2 test with Yates's continuity correction, and with a two-sided significance level of 5%.
Time Frame: 24 hours after the end of surgery
Measure: Count of Participants; unit: Participants
Groups:
- APD421 at 5mg: A 5mg (2mL) dose of APD421 given by slow intravenous (IV) push over one minute at induction of anaesthesia
- Placebo: A 2mL dose of placebo given by slow intravenous (IV) push over one minute at induction of anaesthesia
Arm/Group | APD421 at 5mg | Placebo
Number analyzed (Participants) | 176 | 166
Participants | 78 | 54
Statistical Analysis 1: Comparison: APD421 at 5mg vs Placebo; Test type: Superiority; p = 0.033, Chi-squared, Corrected — 2-sided; Yates's continuity correction

2. Secondary Outcome: Number of Participants With no Nausea.
Description: Nausea (defined as the desire to vomit without the presence of expulsive muscular movements) measured on a 0-10 verbal response scale, where 0=no nausea at all and 10=the worst nausea imaginable. "No nausea" means no score ≥ 1.
Time Frame: 24 hours after end of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | APD421 at 5mg | Placebo
Number analyzed (Participants) | 176 | 166
Participants | 82 | 64
Statistical Analysis 1: Comparison: APD421 at 5mg vs Placebo; Test type: Superiority; p = 0.16, Chi-squared, Corrected; Yates's continuity correction

3. Secondary Outcome: Number of Participants With no Emesis
Description: Emesis is defined as vomiting (production of even the smallest amount of stomach contents) or retching (muscular movements of vomiting but without expulsion of stomach contents, usually because of an empty stomach)
Time Frame: 24 hours after end of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | APD421 at 5mg | Placebo
Number analyzed (Participants) | 176 | 166
Participants | 141 | 129
Statistical Analysis 1: Comparison: APD421 at 5mg vs Placebo; Test type: Superiority; p = 0.68, Chi-squared, Corrected; Yates's continuity correction

4. Secondary Outcome: Number of Participants With no Use of Rescue Medication
Description: Any agent given in the post-operative period with the intention of providing anti-emetic rescue was counted as rescue anti-emetic medication for the purposes of efficacy determination, even if it did not achieve control of emesis or was given incorrectly (e.g., wrong dosage or route). Any agent given in the post-operative period which would be expected, by virtue of its pharmacology, dosage and route, to exert a clinically meaningful anti-emetic effect was considered as rescue anti-emetic medication, even if administered inadvertently or without the intention of providing rescue.
Time Frame: 24 hours after end of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | APD421 at 5mg | Placebo
Number analyzed (Participants) | 176 | 166
Participants | 80 | 55
Statistical Analysis 1: Comparison: APD421 at 5mg vs Placebo; Test type: Superiority; p = 0.026, Chi-squared, Corrected; Yates's continuity correction

5. Secondary Outcome: The Number of Participants With no Emesis, no Significant Nausea and no Use of Rescue Medication
Description: No occurrence of vomiting/retching, no nausea score ≥ 4 on verbal response scale (where 0=no nausea at all and 10=the worst nausea imaginable) and no use of rescue medication.
Time Frame: 24 hours after the end of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | APD421 at 5mg | Placebo
Number analyzed (Participants) | 176 | 166
Participants | 73 | 53
Statistical Analysis 1: Comparison: APD421 at 5mg vs Placebo; Test type: Superiority; p = 0.086, Chi-squared, Corrected; Yates's continuity correction

6. Secondary Outcome: The Number of Participants With no Significant Nausea
Description: Nausea (defined as the desire to vomit without the presence of expulsive muscular movements) measured on a 0-10 verbal response scale, where 0=no nausea at all and 10=the worst nausea imaginable. "No significant nausea" means no score ≥ 4.
Time Frame: 24 hours after the end of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | APD421 at 5mg | Placebo
Number analyzed (Participants) | 176 | 166
Participants | 107 | 84
Statistical Analysis 1: Comparison: APD421 at 5mg vs Placebo; Test type: Superiority; p = 0.074, Chi-squared, Corrected; Yates's continuity correction

7. Secondary Outcome: Number of Participants With "Total Response"
Description: Total response is defined as no occurrence of vomiting/retching, no nausea score ≥ 1 and no use of rescue medication.
Time Frame: 24 hours after the end of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | APD421 at 5mg | Placebo
Number analyzed (Participants) | 176 | 166
Participants | 67 | 50
Statistical Analysis 1: Comparison: APD421 at 5mg vs Placebo; Test type: Superiority; p = 0.15, Chi-squared, Corrected; Yates's continuity correction

ADVERSE EVENTS:
Time Frame: 7 days
Groups:
- APD421 5mg Dose: A 5mg dose of APD421 given by slow push, single intravenous (IV) administration over a time frame of one minute at induction of anaesthesia
- Placebo: Placebo given by single intravenous (IV) administration by slow push over one minute at induction of anaesthesia
Arm/Group | APD421 5mg Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/176 | 0/166
Serious Adverse Events (participants affected / at risk) | 8/176 | 9/166
Other Adverse Events (participants affected / at risk) | 169/176 | 160/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APD421 5mg Dose (N=176) | Placebo (N=166)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anaemia Postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post Procedural Constipation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post Operative Ileus (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APD421 5mg Dose (N=176) | Placebo (N=166)
Anaemia Postoperative (Injury, poisoning and procedural complications) | 31 (31) | 32 (32)
Procedural Pain (Injury, poisoning and procedural complications) | 42 (42) | 41 (41)
Hyperglycaemia (Metabolism and nutrition disorders) | 33 (33) | 38 (38)
Hypocalcaemia (Metabolism and nutrition disorders) | 26 (26) | 30 (30)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 11 (11) | 11 (11)
Hypoproteinaemia (Metabolism and nutrition disorders) | 26 (26) | 25 (25)
Constipation (Gastrointestinal disorders) | 12 (12) | 15 (15)
Abdominal distension (Gastrointestinal disorders) | 12 (12) | 9 (9)
Bood Prolactin Increased (Investigations) | 9 (9) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 12 (12) | 9 (9)

LIMITATIONS AND CAVEATS:
There were no limitations and caveats in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days